CLINICAL TRIAL: NCT01459458
Title: Family Planning-based Partner Abuse Intervention to Reduce Unintended Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elizabeth Miller, Chief of Adolescent Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11050458; NICHD (Other Grant/Funding Number: 1R01HD064407-01A1)
Record Dates: First submitted 2011-10-10; First posted 2011-10-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Violence; Pregnancy
Keywords: intimate partner violence; gender-based violence; domestic violence; unintended pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinics trained in brief intervention (Experimental): Female clients ages 16-29 seeking care in 11 reproductive health clinics in Western Pennsylvania where clinic providers are trained to implement the brief partner violence/reproductive coercion intervention.
  Interventions: Behavioral: Family Planning-based Partner Violence Intervention
- Control sites providing standard of care (No Intervention): Female clients ages 16-29 seeking care in 14 reproductive health clinics in Western Pennsylvania where clinic providers are providing standard domestic violence screening per usual standard of care.

INTERVENTIONS:
Behavioral: Family Planning-based Partner Violence Intervention — The intervention includes three major components:
  1. Enhanced Screening and Education: scripted questions to assess for reproductive coercion and pregnancy risk combined with intimate partner violence (IPV) assessment and education regarding how IPV may affect women's reproductive health with the assistance of a safety/educational card created for this intervention.
  2. Harm Reduction Counseling: assisting clients in identifying and planning strategies to reduce their risk for future unintended pregnancies and IPV.
  3. Supported Referral: educating all clients regarding local resources for victims of IPV and problem-solving regarding barriers to acquisition of these resources as needed.
  Arms: Clinics trained in brief intervention

SUMMARY:
This is a community-based participatory study to test a brief intervention to reduce risk for intimate partner violence (IPV) and associated unintended pregnancy among young, medically underserved women attending family planning (FP) clinics. Women ages 16-29 years utilizing FP clinics report higher rates of IPV compared to their same-age peers, experiences associated with unintended pregnancy. A critical mechanism connecting IPV with poor reproductive health is abusive partners' control of women's reproduction through condom refusal, pressuring women to get pregnant, and birth control sabotage, a phenomenon described as reproductive coercion. In the investigative team's pilot intervention study 53% of young women using FP clinics reported ever experiencing IPV, and 25% reported reproductive coercion, the combination of which was strongly associated with unintended pregnancy. The proposed reproductive coercion/partner violence intervention was developed collaboratively by community-based practitioners, advocates, and researchers, with significant input from FP clients. Designed to be implemented within routine FP care, maximizing feasibility and sustainability of this program, the intervention provides 1) client education and assessment regarding IPV and reproductive coercion; 2) discussion of harm reduction behaviors to reduce risk for unintended pregnancy and IPV victimization, and 3) supported referrals to IPV victim services. This is a full-scale RCT to assess the effects of this innovative program on IPV, reproductive coercion and unintended pregnancy, major health threats for medically underserved women. Evaluation of this intervention will involve random assignment of 25 FP clinics (unit of randomization) in Western PA to either intervention or control (i.e., standard-of-care) conditions. Female FP clients ages 16-29 (N=3600) will be assessed at baseline, 12-20 weeks (FU1), and 12 months (FU2) to assess intervention effects on knowledge and behaviors related to IPV, reproductive coercion and related harm reduction, as well as unintended pregnancy. Data will be collected via audio computer-assisted self-interview in English or Spanish. Chart extraction will track clinic utilization, pregnancy testing, and diagnosed pregnancies. Regression models appropriate for longitudinal data from cluster-randomized trials will be used to estimate intervention effects.

ELIGIBILITY:
Inclusion:

* female clients
* ages 16-29
* English or Spanish speaking
* able to provide their own consent
* plan to be in area for the next 12 months
* willing to be contacted for follow up survey and able to provide additional contact information

Exclusion Criteria:

* female clients not of the specified age range
* neither English nor Spanish speaking
* clients who are intoxicated or otherwise not able to provide their own consent

Ages: 16 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3687 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in partner violence victimization (summary score) | baseline to 12 months
  baseline-adjusted differences in post-intervention partner violence victimization up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}
Change in reproductive coercion (summary score) | baseline to12 months
  baseline-adjusted differences in post-intervention levels of reproductive coercion up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}

SECONDARY OUTCOMES:
Unintended pregnancy | 12 months
  incidence of unintended pregnancy
Change in recognition of abusive behaviors (mean score) | baseline to 12 months
  baseline-adjusted differences in mean post-intervention levels of recognition of what constitutes abusive behavior up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}
Change in harm reduction self-efficacy (mean score) | baseline to 12 months
  baseline-adjusted differences in mean post-intervention levels of self-efficacy regarding uptake of harm reduction strategies up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}
Knowledge regarding violence victimization resources | up to 12 months
  post-intervention levels of knowledge about violence victimization related resources up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}
Harm reduction strategies uptake (summary score) | up to 12 months
  post-intervention levels of uptake of harm reduction strategies up to 12 months {pooled analysis of FU 1 (12-20 weeks) and FU 2 (12 month) score}

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, M.D., Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Pennsylvania Family Planning Clinics, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kalra N, Hooker L, Reisenhofer S, Di Tanna GL, Garcia-Moreno C. Training healthcare providers to respond to intimate partner violence against women. Cochrane Database Syst Rev. 2021 May 31;5(5):CD012423. doi: 10.1002/14651858.CD012423.pub2. PMID 34057734
- [Derived] Hill AL, Miller E, Borrero S, Zelazny S, Miller-Walfish S, Talis J, Switzer GE, Abebe KZ, Chang JC. Family Planning Providers' Assessment of Intimate Partner Violence and Substance Use. J Womens Health (Larchmt). 2021 Sep;30(9):1225-1232. doi: 10.1089/jwh.2020.8699. Epub 2021 Jan 18. PMID 33464993
- [Derived] Miller E, Tancredi DJ, Decker MR, McCauley HL, Jones KA, Anderson H, James L, Silverman JG. A family planning clinic-based intervention to address reproductive coercion: a cluster randomized controlled trial. Contraception. 2016 Jul;94(1):58-67. doi: 10.1016/j.contraception.2016.02.009. Epub 2016 Feb 15. PMID 26892333
- [Derived] Tancredi DJ, Silverman JG, Decker MR, McCauley HL, Anderson HA, Jones KA, Ciaravino S, Hicks A, Raible C, Zelazny S, James L, Miller E. Cluster randomized controlled trial protocol: addressing reproductive coercion in health settings (ARCHES). BMC Womens Health. 2015 Aug 6;15:57. doi: 10.1186/s12905-015-0216-z. PMID 26245752
- [Derived] Miller E, McCauley HL, Tancredi DJ, Decker MR, Anderson H, Silverman JG. Recent reproductive coercion and unintended pregnancy among female family planning clients. Contraception. 2014 Feb;89(2):122-8. doi: 10.1016/j.contraception.2013.10.011. Epub 2013 Dec 10. PMID 24331859